CLINICAL TRIAL: NCT02116972
Title: A Double-Blind, Randomized, Parallel Group, Dose-Ranging Study to Assess the Safety and Efficacy of FX006 for the Treatment of Pain in Patients With Osteoarthritis of the Knee
Brief Title: Study of FX006 vs Normal Saline in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX006-2014-006
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; pain; corticosteroid; intra-articular; injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — FX006; Triamcinolone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- FX006 16 mg (Experimental): Single 5 mL intra-articular (IA) injection Extended-release formulation
  Interventions: Drug: FX006 16 mg
- FX006 32 mg (Experimental): Single 5 mL intra-articular (IA) injection Extended-release formulation
  Interventions: Drug: FX006 32 mg
- Placebo (Placebo Comparator): Normal Saline Single 5 mL intra-articular (IA) injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FX006 32 mg — Single 5 mL IA injection
  Other Names: Zilretta
  Arms: FX006 32 mg
Drug: Placebo — Single 5 mL IA injection
  Other Names: Normal Saline
  Arms: Placebo
Drug: FX006 16 mg — Single 5 mL IA injection
  Arms: FX006 16 mg

SUMMARY:
The purpose of this study was to assess the magnitude and duration of pain relief of a single IA injection of 2 doses (16 and 32 mg) of FX006, an extended-release formulation of TCA, relative to normal saline (placebo control).

DETAILED DESCRIPTION:
This was a double-blind, randomized, parallel group, dose-ranging, single-dose study. The study was conducted in male and female patients ≥40 years of age with OA of the knee.

Approximately 300 patients with OA of the knee were randomized, using a centralized randomization procedure, to 1 of 3 treatment groups (1:1:1) and treated with a single IA injection of:

* 16 mg FX006,
* 32 mg FX006, or
* normal saline (placebo).

Each patient was evaluated for a total of 24 weeks following a single IA injection. Following screening, safety and efficacy were evaluated at 7 out-patient visits (Days 1 [Baseline], Weeks 4, 8, 12, 16, 20, and 24).

The study was expected to enroll over approximately 6 to 7 months.

ELIGIBILITY:
Main Inclusion Criteria:

* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Male or female >=40 years of age
* Has documented diagnosis of OA of the index knee made at least 6 months prior to Screening
* Currently meets American College of Rheumatology (ACR) Criteria (clinical and radiological) for OA
* Kellgren-Lawrence (K-L) Grade 2 or 3 in the index knee per Screening X-ray
* Qualifying mean score on the 24-h average pain score (0-10 numeric rating scale)
* Body mass index (BMI) ≤ 40 kg/m2
* Willingness to abstain from use of restricted medications

Main Exclusion Criteria:

* Ipsilateral hip OA
* Fibromyalgia, chronic pain syndrome or other concurrent medical or arthritic conditions which could interfere with the evaluation of the index knee
* History of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis or amyloidosis
* History of arthritides due to crystals (e.g., gout, pseudogout)
* History or clinical signs and symptoms of infection in the index joint
* Knee pain that is not clinically attributable to OA of the knee (e.g., radicular low back pain and hip pain that is referred to the knee that could cause misclassification)
* Pain in any other area of the lower extremities or back that is equal to or greater than the index knee pain
* IA corticosteroid (investigational or marketed) in any joint within 3 months of Screening
* IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
* Intramuscular (IM) corticosteroids (investigational or marketed) within 3 months of Screening
* Oral corticosteroids (investigational or marketed) within 1 month of Screening
* Inhaled, intranasal and topical corticosteroids (investigational or marketed) within 2 weeks of Screening
* Any other IA investigational drug/biologic within 6 months of Screening
* Prior use of FX006
* Women of child-bearing potential not using effective contraception or who are pregnant or nursing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bodick, MD, Study Director — Flexion Therapeutics
Locations (44):
- United States (39):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Anaheim, California
  - Canoga Park, California
  - El Cajon, California
  - Los Angeles, California
  - North Hollywood, California
  - San Diego, California
  - Stamford, Connecticut
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Orlando, Florida
  - Pinellas Park, Florida
  - Tampa, Florida
  - Marietta, Georgia
  - Evansville, Indiana
  - Paducah, Kentucky
  - Wheaton, Maryland
  - New Bedford, Massachusetts
  - Troy, Michigan
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - New York, New York
  - Rochester, New York
  - Raleigh, North Carolina
  - Oklahoma City, Oklahoma
  - Altoona, Pennsylvania
  - Duncansville, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Victoria, Texas
  - Danville, Virginia
- Canada (5):
  - Kitchener, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Québec

REFERENCES:
- [Derived] Conaghan PG, Cohen SB, Berenbaum F, Lufkin J, Johnson JR, Bodick N. Brief Report: A Phase IIb Trial of a Novel Extended-Release Microsphere Formulation of Triamcinolone Acetonide for Intraarticular Injection in Knee Osteoarthritis. Arthritis Rheumatol. 2018 Feb;70(2):204-211. doi: 10.1002/art.40364. Epub 2017 Dec 20. PMID 29088579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for study eligibility at 48 study centers in the United States (US) and Canada. Enrollment took approximately 7 months.
Pre-assignment Details: Subjects were screened within 21 days of being randomized
Groups:
- FX006 16 mg: 102 subjects received FX006 16 mg a single 5 mL IA injection
- FX006 32 mg: 104 subjects received FX006 32 mg a single 5 mL IA injection
- Placebo: 100 subjects received normal saline as a single 5 mL IA injection
Period: Overall Study
Arm/Group | FX006 16 mg | FX006 32 mg | Placebo
Started | 102 | 104 | 104
Completed | 83 | 87 | 85
Not Completed | 19 | 17 | 19
Not completed — Adverse Event | 4 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 5
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Lost to Follow-up | 4 | 3 | 1
Not completed — Lack of Efficacy | 6 | 6 | 5
Not completed — scheduling conflicts and relocation | 3 | 3 | 6

BASELINE CHARACTERISTICS:
Population: A total of 310 subjects were randomized to a treatment assignment but only 306 enrolled subjects received their randomized treatment. Four (4) subjects randomized to placebo arm were were not treated.
Groups:
- FX006 16 mg; FX006 32 mg: Single intra-articular injection
  FX006: Single intra-articular injection
- Normal Saline: Single intra-articular injection
  Normal saline: Single intra-articular injection
- Total: Total of all reporting groups
Arm/Group | FX006 16 mg | FX006 32 mg | Normal Saline | Total
Number analyzed (Participants) | 102 | 104 | 100 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (8.34) | 58.7 (8.06) | 59.7 (8.23) | 58.8 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 51 | 61 | 174
  Male | 40 | 53 | 39 | 132

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Weekly Mean of the Average Daily (24-hr) Pain Intensity Scores for 32 mg FX006 Versus Placebo
Description: The pain intensity score is measured using an 11-point numeric rating scale (NRS), where 0 indicates "no pain"and 10 indicates "pain as bad as you can imagine."
Time Frame: Baseline and Week 12
Population: Randomized patients who received study drug assigned to the FX006 32 mg arm and the placebo arm
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- FX006 32 mg: FX006: Single 5 mL IA injection
- Placebo: Normal Saline: Single 5 mL IA injection
Arm/Group | FX006 32 mg | Placebo
Number analyzed (Participants) | 104 | 100
units on a scale | -3.08 (0.229) | -2.50 (0.238)
Statistical Analysis 1: Comparison: FX006 32 mg vs Placebo; The step-down testing procedure to control for multiplicity would be voided if the primary endpoint is not met and analyses proceeded for exploratory purposes; Test type: Superiority; p = 0.0821, Logitudinal mixed effects model; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.22 to 0.07]

2. Secondary Outcome: Change From Baseline to Week 12 for WOMAC C (Function Subscale)
Description: The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo
Number analyzed (Participants) | 104 | 100
units on a scale | -1.01 (0.083) | -0.79 (0.087)

3. Secondary Outcome: Change From Baseline to Week 12 for Patient Global Impression of Change (PGIC)
Description: The Patient Global Impression of Change is a scale that aims to evaluate all aspects of participants' (patients') health and determining if there has been an improvement or not. The participant selects the one response from the response options that gives the most accurate description of his/her state of health (overall status). This is a 7-point scale, and scores range from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores indicate better health status.
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo
Number analyzed (Participants) | 104 | 100
units on a scale | 2.6 (0.14) | 2.7 (0.14)

4. Secondary Outcome: Change From Baseline to Week 16 and Then Week 20 and Then Week 24 in the Weekly Mean of the Average Daily (24-hour) Pain Intensity Scores
Description: The pain intensity score is measured using an 11-point numeric rating scale (NRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine."
Time Frame: Baseline and Weeks 16, 20 and 24
Population: Randomized patients who received study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo
Number analyzed (Participants) | 104 | 100
units on a scale
  Week 16: number analyzed (Participants) | 97 | 86
  Week 16 | -2.83 (0.2224) | -2.46 (0.234)
  Week 20: number analyzed (Participants) | 91 | 82
  Week 20 | -2.81 (0.233) | -2.34 (0.244)
  Week 24: number analyzed (Participants) | 78 | 68
  Week 24 | -2.51 (0.241) | -2.24 (0.252)

5. Other Pre Specified Outcome: Percent of Responders According to Outcomes Measures in OMERACT-OARSI Strict Criteria
Description: Outcome Measures in Rheumatoid Arthritis Clinical Trials - Osteoarthritis Research Society International. (OMERACT-OARSI) Responders are defined as participants with high improvement in pain or function.
Time Frame: Weeks 4, 8 and 12
Population: Percent of responders according to Outcomes Measures in OMERACT-OARSI strict criteria for patients assigned to FX006 16 mg arm was not a pre-specified Secondary Outcome and therefore not reported.
Measure: Count of Participants; unit: Participants
Arm/Group | FX006 32 mg | Placebo
Number analyzed (Participants) | 104 | 100
Participants
  Week 4: number analyzed (Participants) | 104 | 98
  Week 4 | 75 | 51
  Week 8: number analyzed (Participants) | 104 | 94
  Week 8 | 73 | 58
  Week 12: number analyzed (Participants) | 101 | 92
  Week 12 | 70 | 57

6. Other Pre Specified Outcome: Change From Baseline to Week 12 for WOMAC C (Function Subscale)
Description: The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5- point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- FX006 16 mg: FX006: Single 5 mL IA injection
Arm/Group | FX006 16 mg | Placebo
Number analyzed (Participants) | 102 | 100
units on a scale | -0.83 (0.085) | -0.79 (0.087)

7. Other Pre Specified Outcome: Change From Baseline to Week 12 for Patient Global Impression of Change (PGIC)
Description: as for outcome 3
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 16 mg | Placebo
Number analyzed (Participants) | 102 | 100
units on a scale | 2.5 (0.14) | 2.7 (0.14)

8. Other Pre Specified Outcome: Change From Baseline to Each Week in Weekly Mean of the ADP Intensity Scores
Description: The pain intensity score is measured using an 11-point numeric rating scale (NRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine."Weeks 12, 16, 20, and 24 are specified as the primary and secondary endpoints for the 32 mg group and the placebo group
Time Frame: Baseline and Up to Week 24
Population: Randomized patients who received study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 16 mg | FX006 32 mg | Placebo
Number analyzed (Participants) | 102 | 104 | 100
units on a scale
  Week 1: number analyzed (Participants) | 100 | 103 | 100
  Week 1 | -2.04 (0.177) | -1.96 (0.175) | -1.24 (0.178)
  Week 2: number analyzed (Participants) | 101 | 103 | 99
  Week 2 | -2.88 (0.218) | -2.75 (0.216) | -1.65 (0.220)
  Week 3: number analyzed (Participants) | 100 | 103 | 94
  Week 3 | -2.90 (0.228) | -2.91 (0.226) | -1.74 (0.231)
  Week 4: number analyzed (Participants) | 98 | 101 | 93
  Week 4 | -3.05 (0.228) | -3.20 (0.226) | -1.84 (0.232)
  Week 5: number analyzed (Participants) | 97 | 100 | 93
  Week 5 | -3.28 (0.222) | -3.39 (0.219) | -2.05 (0.225)
  Week 6: number analyzed (Participants) | 97 | 101 | 91
  Week 6 | -3.27 (0.225) | -3.29 (0.222) | -2.20 (0.229)
  Week 7: number analyzed (Participants) | 97 | 102 | 92
  Week 7 | -3.14 (0.233) | -3.13 (0.230) | -2.28 (0.237)
  Week 8: number analyzed (Participants) | 95 | 101 | 91
  Week 8 | -3.08 (0.237) | -3.04 (0.234) | -2.33 (0.242)
  Week 9: number analyzed (Participants) | 91 | 98 | 92
  Week 9 | -3.09 (0.233) | -3.24 (0.229) | -2.39 (0.237)
  Week 10: number analyzed (Participants) | 92 | 98 | 90
  Week 10 | -2.88 (0.229) | -3.17 (0.224) | -2.44 (0.233)
  Week 11: number analyzed (Participants) | 90 | 96 | 90
  Week 11 | -2.78 (0.234) | -3.18 (0.229) | -2.48 (0.238)
  Week 12: number analyzed (Participants) | 90 | 96 | 89
  Week 12 | -2.59 (0.234) | -3.08 (0.229) | -2.50 (0.238)
  Week 13: number analyzed (Participants) | 90 | 96 | 88
  Week 13 | -2.68 (0.234) | -3.12 (0.229) | -2.43 (0.239)
  Week 14: number analyzed (Participants) | 89 | 96 | 85
  Week 14 | -2.38 (0.235) | -2.83 (0.229) | -2.48 (0.239)
  Week 15: number analyzed (Participants) | 86 | 95 | 88
  Week 15 | -2.38 (0.225) | -2.91 (0.219) | -2.44 (0.229)
  Week 16: number analyzed (Participants) | 87 | 97 | 86
  Week 16 | -2.30 (0.231) | -2.83 (0.224) | -2.46 (0.234)
  Week 17: number analyzed (Participants) | 82 | 96 | 88
  Week 17 | -2.32 (0.237) | -2.71 (0.229) | -2.41 (0.240)
  Week 18: number analyzed (Participants) | 82 | 91 | 86
  Week 18 | -2.32 (0.240) | -2.73 (0.232) | -2.34 (0.242)
  Week 19: number analyzed (Participants) | 82 | 91 | 85
  Week 19 | -2.27 (0.241) | -2.76 (0.233) | -2.28 (0.243)
  Week 20: number analyzed (Participants) | 81 | 91 | 82
  Week 20 | -2.27 (0.241) | -2.81 (0.233) | -2.34 (0.244)
  Week 21: number analyzed (Participants) | 76 | 85 | 76
  Week 21 | -2.21 (0.246) | -2.71 (0.237) | -2.38 (0.248)
  Week 22: number analyzed (Participants) | 72 | 81 | 71
  Week 22 | -2.41 (0.249) | -2.53 (0.240) | -2.30 (0.251)
  Week 23: number analyzed (Participants) | 72 | 78 | 71
  Week 23 | -2.33 (0.258) | -2.40 (0.249) | -2.25 (0.260)
  Week 24: number analyzed (Participants) | 71 | 78 | 68
  Week 24 | -2.38 (0.249) | -2.51 (0.241) | -2.24 (0.252)

9. Other Pre Specified Outcome: Change From Baseline to Each of Weeks 4, 8, 16, 20, and 24 in WOMAC-C-function
Description: as for outcome 2
Time Frame: Baseline and Weeks 4, 8, 16, 20 and 24 (Week 12 data is represented in the secondary outcome measure)
Population: Change from baseline to each of Weeks 4, 8, 16, 20, and 24 in WOMAC-C-function for patients assigned to FX006 16 mg arm was not a pre-specified Secondary Outcome and therefore not reported
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo
Number analyzed (Participants) | 104 | 100
units on a scale
  Week 4: number analyzed (Participants) | 104 | 95
  Week 4 | -1.16 (0.079) | -0.66 (0.082)
  Week 8: number analyzed (Participants) | 103 | 93
  Week 8 | -1.09 (0.082) | -0.74 (0.085)
  Week 16: number analyzed (Participants) | 95 | 87
  Week 16 | -0.94 (0.083) | -0.84 (0.086)
  Week 20: number analyzed (Participants) | 92 | 87
  Week 20 | -0.87 (0.082) | -0.84 (0.085)
  Week 24: number analyzed (Participants) | 80 | 76
  Week 24 | -0.89 (0.083) | -0.80 (0.086)

10. Other Pre Specified Outcome: Change From Baseline to Each of Weeks 4, 8, 12, 16, 20, and 24 in WOMAC-A Pain
Description: as for outcome 2
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 24
Population: Change from baseline to each of Weeks 4, 8, 12, 16, 20, and 24 in WOMAC-A pain for patients assigned to FX006 16 mg arm was not a pre-specified Secondary Outcome and therefore not reported.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo
Number analyzed (Participants) | 104 | 100
units on a scale
  Week 4: number analyzed (Participants) | 104 | 95
  Week 4 | -1.11 (0.080) | -0.64 (0.082)
  Week 8: number analyzed (Participants) | 104 | 93
  Week 8 | -1.09 (0.083) | -0.71 (0.087)
  Week 12: number analyzed (Participants) | 100 | 90
  Week 12 | -0.98 (0.080) | -0.81 (0.083)
  Week 16: number analyzed (Participants) | 95 | 87
  Week 16 | -0.95 (0.083) | -0.80 (0.087)
  Week 20: number analyzed (Participants) | 92 | 87
  Week 20 | -0.89 (0.083) | -0.84 (0.086)
  Week 24: number analyzed (Participants) | 80 | 76
  Week 24 | -0.91 (0.084) | -0.78 (0.086)

11. Other Pre Specified Outcome: Change From Baseline to Each of Weeks 4, 8, 16, 20, and 24 in PGIC
Description: as for outcome 3
Time Frame: Baseline and Weeks 4, 8, 16, 20, and 24 (Week 12 data reported in secondary outcome measure)
Population: Change from baseline to each of Weeks 4, 8, 16, 20, and 24 in PGIC for patients assigned to FX006 16 mg arm was not a pre-specified Secondary Outcome and therefore not reported.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 32 mg | Placebo
Number analyzed (Participants) | 104 | 100
units on a scale
  Week 4: number analyzed (Participants) | 104 | 94
  Week 4 | 2.2 (0.13) | 3.0 (0.13)
  Week 8: number analyzed (Participants) | 104 | 93
  Week 8 | 2.4 (0.14) | 2.8 (0.14)
  Week 16: number analyzed (Participants) | 95 | 87
  Week 16 | 2.8 (0.16) | 2.7 (0.16)
  Week 20: number analyzed (Participants) | 92 | 87
  Week 20 | 2.9 (0.15) | 2.8 (0.16)
  Week 24: number analyzed (Participants) | 80 | 76
  Week 24 | 2.7 (0.16) | 3.1 (0.16)

12. Other Pre Specified Outcome: Proportion of Patients Experiencing a >20%, 30% and 50% Decrease in Pain From Baseline in Weekly Mean of the Average Daily (24-hr) Pain Intensity Scores at Week 12
Description: as for outcome 4
Time Frame: 12 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Time to Onset of Pain Relief
Description: Time to onset of pain relief in days is defined as the time from administration of study treatment to the first pain assessment showing >30% improvement from the weekly average daily pain score at baseline.
Time Frame: Baseline up to 24 Weeks after administration of study treatment
Population: Time to onset of pain relief for patients assigned to FX006 16 mg arm was not a pre-specified Secondary Outcome and therefore not reported.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FX006 32 mg | Placebo
Number analyzed (Participants) | 104 | 100
days | 4 [3 to 8] | 8 [5 to 17]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected following IA administration through the final study visit.
Description: A total of 310 subjects were randomized to a treatment assignment but only 306 enrolled subjects received their randomized treatment. Four (4) subjects randomized to placebo arm were were not treated.
Arm/Group | FX006 16 mg | FX006 32 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/104 | 0/100
Serious Adverse Events (participants affected / at risk) | 1/102 | 3/104 | 0/100
Other Adverse Events (participants affected / at risk) | 14/102 | 13/104 | 21/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 16 mg (N=102) | FX006 32 mg (N=104) | Placebo (N=100)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 16 mg (N=102) | FX006 32 mg (N=104) | Placebo (N=100)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 8 (8) | 16 (16)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 5 (5)

LIMITATIONS AND CAVEATS:
Subsequent to completion of clinical studies extensive testing was performed to assess the actual dose delivered. It was determined that the FX006 delivered dose to the patient from an FX006 40 mg vial is 32 mg and from FX006 20 mg vial is 16 mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes